CLINICAL TRIAL: NCT06339047
Title: The Effect of Projector Kaleidoscope and Cartoons in the Operating Room on Anxiety, Fear and Pain in Children Aged 4-10 Who Will Undergo Outpatient Surgery
Brief Title: The Effect of Projector Kaleidoscope and Cartoons on Anxiety, Fear, and Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/09
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Anxiety and Fear; Pain; Surgery
Keywords: anxiety; fear; pain; day surgery
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Projector Kaleidoscope (Experimental): Children in the projector kaleidoscope group will be watched for approximately 5 minutes before induction into the operating room.
  Interventions: Other: Projector Kaleidoscope
- Cartoon (Experimental): Children in the cartoon group will be asked which cartoon they want to watch from the cartoon pool and will be shown the cartoon they want. The cartoon duration is approximately 5 minutes.
  Interventions: Other: Cartoon
- Control (No Intervention): Routine care will be given

INTERVENTIONS:
Other: Projector Kaleidoscope — Children in the projector kaleidoscope group will be watched for approximately 5 minutes before induction in the operating room.
  Arms: Projector Kaleidoscope
Other: Cartoon — Children in the cartoon group will be asked which cartoon they want to watch from the cartoon pool and will be shown the cartoon they want. The cartoon duration is approximately 5 minutes.
  Arms: Cartoon

SUMMARY:
The research will be conducted with children hospitalized in Tarsus State Hospital Children's Clinics and who meet the sampling criteria.

The population of the study, which is planned as a randomized controlled experimental study, will consist of children aged 4-10 years old who are admitted to the pediatric surgery service of Tarsus State Hospital and will undergo outpatient surgical intervention.

In collecting research data; the Introductory Information Form, Child Anxiety Scale, Child Fear Scale, Wong-Baker Pain Scale and Vital Signs Follow-up Form will be used.

DETAILED DESCRIPTION:
The research will be conducted with children hospitalized in Tarsus State Hospital Children's Clinics and who meet the sampling criteria.

The population of the study, which is planned as a randomized controlled experimental study, will consist of children aged 4-10 years old who are admitted to the pediatric surgery service of Tarsus State Hospital and will undergo outpatient surgical intervention.

In collecting research data; the Introductory Information Form, Child Anxiety Scale, Child Fear Scale, Wong-Baker Pain Scale, and Vital Signs Follow-up Form will be used.

Collection of Data The research will be implemented after ethics committee approval and written institutional permission are obtained.

Stage 1: By consulting experts on the subject, the researchers will create a pool of cartoons suitable for the level of children in the 4-10 age group that they can watch. The created children's cartoon pool will be sent to people who are experts in the field (child development specialists, child psychiatrists, and pediatric nurses).

Stage 2: Data collection forms to be used before the research. A pilot study will be conducted with 10 children to evaluate the suitability of the cartoon for children.

Stage 3: The children and their parents in the sample group will be informed about the method followed in the application and the research, and their verbal and written permissions will be obtained.

Stage 4: The introductory information form in the research will be applied to the children in the sample group.

Stage 5: Randomization will be achieved by randomly and equally distributing patients who meet the sample selection criteria to 3 groups (1st experimental group, 2nd experimental control group and 3rd group control group) through a computer program.

(http://www1.assumption.edu/users/avadum/applets/RandAssign/GroupGen.html). Stage 6: Children in the projector kaleidoscope group will be watched for approximately 5 minutes before induction in the operating room. Children in the cartoon group will be asked which cartoon they want to watch from the cartoon pool and will be shown the cartoon they want. The cartoon duration is approximately 5 minutes.

Stage 7: Before the surgery, the anxiety, fear and vital signs of the children in the sample will be evaluated. Children's fear assessment will be done by both the child and the nurse. Since parents are not allowed into the operating room, the evaluation will be made only by the child and the nurse.

Stage 8: In the postoperative period, the anxiety, fear, vital signs and pain of the children in the experimental and control groups will be recorded. Children's fear and pain assessment will be done by the child, nurse and parent.

Analysis of Research Data:

The data obtained in the study were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 25.0 program. Descriptive statistical methods (number, percentage, min-max values, mean, and standard deviation) will be used when evaluating the data. The suitability of the data used for normal distribution will be checked with kurtosis and skewness values. In comparing quantitative data with normally distributed data, an independent t-test will be used for the difference between two independent groups. In comparing more than two dependent groups, analysis of variance will be applied in repeated measurements and in case of a difference, Bonferroni will be used to find the group that makes the difference. In comparing quantitative data in non-normally distributed data, the Mann-Whitney U test will be applied for the difference between two independent groups, and in comparing more than two dependent groups, the Friedman test will be applied, and in case of a difference, the corrected Bonferroni will be used to find the group that makes the difference. Chi-square analysis will be applied to test the relationship between categorical variables. Cohen's Kappa Test will be applied in interobserver agreement analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 4-10
* Having outpatient surgery
* Volunteering to participate in the study

Exclusion Criteria:

* Having had a previous surgical intervention
* Having a chronic disease
* The child has visual, hearing, and mental disabilities

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Anxiety | 1 day
  Child Anxiety Scale-State scale will be used. The scale is shaped like a thermometer with a bulb at the bottom and horizontal lines at intervals going upwards. This scale, for children ages 4 to 10, asks children, "Imagine that all your anxious or nervous emotions are in the bulb or bottom part of the thermometer" or "If you're a little anxious or nervous, the emotions might move up a little bit on the thermometer." If you're very, very anxious or nervous, emotions can run rampant. "Put a line on the thermometer that shows how anxious or angry you are." To measure state anxiety, the child is asked to indicate what he or she is feeling "right now." The score can vary between 0 and 10
Fear | 1 day
  "Children's Fear Scale" will be used. This Scale includes 5 different facial expressions. This scale is scored between 0-4 and is stated to be a reliable and valid measurement tool in the assessment of fear.
Pain after surgery | 1 day
  The Wong-Baker scale will be used. There are six facial expressions scored from zero to five. The Wong-Baker Scale has faces that indicate increasing pain intensity from zero to five from left to right.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus State Hospital, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasnia F, Aghebati N, Miri HH, Etezadpour M. Effects of Patient Education and Distraction Approaches Using Virtual Reality on Pre-operative Anxiety and Post-operative Pain in Patients Undergoing Laparoscopic Cholecystectomy. Pain Manag Nurs. 2023 Jun;24(3):280-288. doi: 10.1016/j.pmn.2022.12.006. Epub 2023 Jan 17. PMID 36658058
- [Background] Atalay, B., Güler, R., & Haylı, Ç.M.(2021). Investıgatıon of preoperatıve anxıety levels ın pedıatrıc groups. Turkish Journal of Health Science and Life, 4(1), 24-26.
- [Background] Baghele A, Dave N, Dias R, Shah H. Effect of preoperative education on anxiety in children undergoing day-care surgery. Indian J Anaesth. 2019 Jul;63(7):565-570. doi: 10.4103/ija.IJA_37_19. PMID 31391620
- [Background] Bartik K, Toruner EK. Effectiveness of a Preoperative Preparation Program on Children's Emotional States and Parental Anxiety. J Perianesth Nurs. 2018 Dec;33(6):972-980. doi: 10.1016/j.jopan.2017.09.008. Epub 2017 Nov 20. PMID 30449445
- [Background] Bülbül, F., &Arıkan B. (2018). Çocuklarda ameliyat öncesi psikolojik hazırlık:Güncel Yaklaşımlar. Balıkesır Health Scıences Journal, 7(3), 101-107.
- [Background] Chartrand J, Tourigny J, MacCormick J. The effect of an educational pre-operative DVD on parents' and children's outcomes after a same-day surgery: a randomized controlled trial. J Adv Nurs. 2017 Mar;73(3):599-611. doi: 10.1111/jan.13161. Epub 2016 Oct 20. PMID 27681601
- [Background] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Background] Ersig, A.L.,Kleiber, C., McCarthy, A.M., ve Hanrahan, K. (2013). Validation of a clinicallyusefulmeasure of children'sstateanxietybeforemedicalprocedures. JournalforSpecialists in PediatricNursing, 18(4), 311-319.
- [Background] Gai N, Naser B, Hanley J, Peliowski A, Hayes J, Aoyama K. A practical guide to acute pain management in children. J Anesth. 2020 Jun;34(3):421-433. doi: 10.1007/s00540-020-02767-x. Epub 2020 Mar 31. PMID 32236681
- [Background] Gerçeker, G. Ö., Ayar, D., Özdemir, Z., & Bektaş, M. (2018). Çocuk anksiyeteskalası-durumluluk ve çocuk Korku ölçeğinin Türk diline kazandırılması. Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 11(1), 9-13.
- [Background] Liu W, Xu R, Jia J, Shen Y, Li W, Bo L. Research Progress on Risk Factors of Preoperative Anxiety in Children: A Scoping Review. Int J Environ Res Public Health. 2022 Aug 9;19(16):9828. doi: 10.3390/ijerph19169828. PMID 36011459
- [Background] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Background] Tadesse, M., Ahmed, S., Regassa, T., Girma, T., Hailu, S., Mohammed, A., &Mohammed, S. (2022). Effect of preoperativeanxiety on postoperativepain on patientsundergoingelectivesurgery: Prospectivecohortstudy. Annals of MedicineandSurgery, 73, 103190
- [Background] Stamenkovic DM, Rancic NK, Latas MB, Neskovic V, Rondovic GM, Wu JD, Cattano D. Preoperative anxiety and implications on postoperative recovery: what can we do to change our history. Minerva Anestesiol. 2018 Nov;84(11):1307-1317. doi: 10.23736/S0375-9393.18.12520-X. Epub 2018 Apr 5. PMID 29624026
- [Background] Yaz, Ş. B.,&Yilmaz, H. B. (2022). Theeffects of designing an educationalanimationmovie in virtualreality on preoperativefearandpostoperativepain in pediatricpatients: A Randomizedcontrolledtrial. Journal of PeriAnesthesiaNursing,37 (3), 357-364